CLINICAL TRIAL: NCT01552590
Title: Effect of Samsca on Control of Hyponatremia and Extracellular Fluid in Cirrhotic Patients With Ascites
Acronym: ECF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 156-KOB-1101i
Record Dates: First submitted 2012-02-21; First posted 2012-03-13 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2014-10

CONDITIONS: Hyponatremia and Extracellular Fluid in Cirrhotic
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Active Comparator): Tablet, QD, 2 weeks
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Tablet, QD, 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan
  Arms: Tolvaptan
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy of a 2-week course of tolvaptan in improving serum sodium and the excretion of extracellular fluid in liver cirrhotic patients with ascites and hyponatremia

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 20 years
2. Subjects who have been diagnosed with hyponatremia [serum sodium < 125 mEq/L or less marked hyponatremia that is symptomatic and has resisted correction with fluid restriction]
3. Subjects who have been diagnosed with an ascites on the abdominal ultrasound.
4. Subjects who have diagnosed with cirrhosis.
5. Subject or their legally acceptable representatives are able to provide informed consent/assent.

Exclusion Criteria:

1. Subject who has ascites by other causes (Tbc, CHF, malignancy, or renal disease) acute severe hyponatemia : Serum Na level < 120 mmol/L and Doubt of symptom caused by hyponatremia and the case which should raise serum Na level urgently based on the investigator's judgment international normalized ratio (INR) >3.0 serum sodium ≥135 mmol/L serum potassium > 5.5 mmol/L Creatinine ≥ 2.0 mg/dL Hepatorenal syndrome defined as 'New International Ascites Club's diagnostic criteria' systolic arterial pressure of < 80 mmHg recent myocardial infarction (< 6 month) spontaneous bacterial peritonitis gastrointestinal bleed ( ≤7 days from randomization) ongoing hepatic encephalopathy of > grade1 known hepatocellular carcinoma intractable ascites
2. Subject who requiring urgent intervention to raise serum sodium acutely
3. Subject who are unable to sense or to respond appropriately to thirst
4. Subject with hypovolemic hyponatremia
5. Subject who should take strong CYP3A inhibitors (clarithromycin, ketoconazole, itraconazole, ritonavir, indinavir, nelfinavir, saquinavir, nefazodone, and telithromycin)
6. Subject who are anuric as no benefit is expected
7. Subject who has genetic defects such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
8. Subject who has fluid depletion
9. Female subjects who are pregnant or lactating
10. Subject judged by the investigator to be inappropriate for inclusion in the trial for any other reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Serum Na | 2 weeks (Baseline, Day 14)

SECONDARY OUTCOMES:
BCM (body composition monitoring) | 7 days
body weight | 7 days
A composite endpoint of ascites worsening | in case
Serum Na normalization rate | 14 days
Biochemistry | 7 days
  Total protein, Albumin, ALP, ALT, AST, r-GT, BUN, Creatinine, Glucose, Cl, K, Na, Ca, Total bilirubin, Uric acid), Hematology (WBC count, Hemoglobin, Hematocrit, Platelets, Serum osm, NT pro-BNP
ECG | 7 days
Adverse event | Daily
Physical examination | 7 days
  HEENT, Thorax, Abdomen, Urogenital, Extremities, Neurological, Skin and Mucosae
Vital signs | Daily
Blood coagulation | 7 days
  PT, INR
Urinalysis | 7 days
  Protein, pH, Glucose, Blood, Bilirubin, Urobilinogen, Random urine Na/K, Urine osm

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Hallym Univ. Chuncheon Sacred Heart Hospital, Bucheon-si
  - Soonchunhyang Univ. Bucheon Hospital, Bucheon-si
  - Wonju Christian Hospital, Wŏnju